CLINICAL TRIAL: NCT05652998
Title: Comparative Study Between Intralesional Injection of Autologous Plasma Rich Platelets Versus Candida Antigen in Patients With Plane Warts
Brief Title: Comparison Between Intralesional Injection of Plasma Rich Platelets and Candida Antigen in Plane Warts
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Randa Abd Al-naser Hussien Kamel, principal investigator, South Valley University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 233/9/21
Record Dates: First submitted 2022-10-27; First posted 2022-12-15 (Actual); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: Plane Wart
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Candida antigen (Active Comparator): patients will be injected with intralesional C.albicans antigen
  Interventions: Biological: C. albicans antigen
- Autologous platelets rich plasma (Active Comparator): patients will receive intralesional autologous PRP injection
  Interventions: Other: autologous PRP
- Saline (Placebo Comparator): patients will receive intralesional saline
  Interventions: Other: saline

INTERVENTIONS:
Biological: C. albicans antigen — a test dose (0.1 ml) of the C. albicans antigen will be injected intradermally into the skin of the forearm. A reaction will be considered positive in presence of ≥5 mm erythema and induration after 48-72 hr. Only reactors will be included. patients will receive intralesional injection of candida antigen at a dose 0.1 ml of 1/1000 solution into the largest wart at 3 weekly intervals for a total of 3 doses.
  Arms: Candida antigen
Other: autologous PRP — patients will receive intralesional autologous PRP injection every month until a complete clearance or for a maximum of 2 sessions. 20 cc blood will be collected under a complete aseptic condition in citrate tubes . The lower 2-4 cc of the plasma will be provided as PRP concentrate after centrifugation. 0.1 ml of PRP will be injected intralesional with an insulin syringe.
  Arms: Autologous platelets rich plasma
Other: saline — patients will receive intralesional saline at a dose of 0.3ml into the largest wart at 2-week intervals until complete clearance is achieved or for a maximum of five treatment
  Arms: Saline

SUMMARY:
To compare the efficacy of intralesional injection of autologous plasma rich platelets and candida antigen in treatment of patients with plane warts .

DETAILED DESCRIPTION:
Cutaneous warts are benign tumors caused by infection of keratinocytes by different serotypes of human papillomavirus(HPV). Its incidence increases during the school years to reach a peak in adolescence and early adulthood, then declines rapidly through the twenties and more gradually thereafter.

Plane warts are mainly caused by HPV serotypes 3, 10, 28, and 41, presenting mainly in children and young adults. They present as skin colored or may be hyperpigmented smooth-surfaced, slightly elevated or flat-topped papules. They are polygonal or round in shape and range in sizes from 1 to 5 mm. The main sites of predilection for the plane warts are the face, dorsal aspects of the hands and forearms, often in a linear array.

Platelet rich plasma (PRP) is an autologous blood-derived product enriched in platelets. Platelets, also called thrombocytes, are blood cells that cause blood clots and other necessary growth healing functions. PRP represents a new bio technology that is part of the growing interest in tissue engineering and cellular therapy today. While it is of autologous origin, it reduces the possibility of adverse effects and transfusion-transmitted infections, so it is well-tolerated therapy for the patients. PRP has been used in the treatment of many cutaneous diseases such as alopecia and acne vulgaris. Its utility has been extended to other cutaneous diseases as melasma, hyperpigmentation, and burns, wherever it elicits tissue repair and regeneration.

Intralesional immunotherapy depends on the ability of the immune system to recognize certain viral, bacterial, and fungal antigens, such as Candida or Trichophyton antigens that induce a delayed-type hypersensitivity reaction, not only to the antigen but also against the wart virus, which in turn increases the ability of the immune system to recognize and eradicate HPV. This stimulated immune response could then subsequently destroy all the injected and noninjected lesions on the body, rather than the locally treated lesion.

Intralesional antigen immunotherapy has recently received increased attention and is considered by many authors a promising modality for the treatment of different types of warts, including the recurrent and recalcitrant variants.

ELIGIBILITY:
Inclusion Criteria:

* Patients proved as having clinically evident plane warts.
* Patients with both sexes with no age limits.

Exclusion Criteria:

* Patient receiving immune suppressive drugs.
* Patients with major comorbidities or concomitant malignancies.
* Patients with any evidence of immunosuppression including HIV infection.
* Patients with any eczematous skin disorder
* Those with any history of hypersensitivity to Candida albicans antigen.
* Patients with chronic systemic medical diseases and bleeding disorders .

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-10-15 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-04-15 (Estimated)

PRIMARY OUTCOMES:
Treatment of plane wart | 6 months
  Evaluation of the efficacy of intradermal injection of candida albicans antigen versus autologous platelet rich plasma in treatment of plane warts

SECONDARY OUTCOMES:
Treatment of plane wart | 6 Months
  Response to treatment will be evaluated by the decrease in size of warts. Lesions with size decrease of less than 50% will be defined as no therapeutic response, size decrease between 50 and 99% as relative response, and complete removal of the lesions will be considered as complete cure.

CONTACTS AND LOCATIONS:
Overall Officials: Hassan M Ibrahim, Ass. Prof., Study Director — Faculty of Medicine - South Valley University; Mohamed A Ali, Prof. Dr., Study Director — Faculty of Medicine - Sohag University; Eisa M Hegazy, Ass. Prof., Study Director — Faculty of Medicine - South Valley University
Locations (1):
- South Valley University, Qina, Egypt